CLINICAL TRIAL: NCT03784742
Title: Investigation of the Effects of Daily Nitrate Consumption on Oral Bacteria Composition, Blood Pressure and Vascular Functio
Brief Title: Effects of Daily Nitrate Consumption on Oral Bacteria Composition, Blood Pressure and Vascular Function
Acronym: REBOC2
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: Saudi Cultural Bureau (Unknown)
Responsible Party: Principal Investigator, Julie Lovegrove, Professor of Human Nutrition, Head of the Hugh Sinclair Unit of Human Nutrition, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: 347890
Record Dates: First submitted 2018-11-01; First posted 2018-12-24 (Actual); Last update posted 2024-04-12 (Actual); Status verified 2024-04

CONDITIONS: No Dental Disease; Non-smoking

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nitrate-rich Beetroot juice (Active Comparator): Nitrate-rich beetroot juice equivalent to 3.7 mg nitrate per kg body weight daily for 8 weeks.
  Interventions: Other: Nitrate rich beetroot juice
- Placebo beetroot juice (Placebo Comparator): Placebo beetroot juice (equivalent volume to the amount of nitrate-rich beetroot juice consumed) daily for 8 weeks.
  Interventions: Other: Placebo beetroot juice

INTERVENTIONS:
Other: Nitrate rich beetroot juice — James White Drinks Limited beetroot juice (0.4-0.45 g nitrate/70 ml drink).
  Arms: Nitrate-rich Beetroot juice
Other: Placebo beetroot juice — James White Drinks Limited Placebo beetroot juice (0 nitrate/70 ml drink).
  Arms: Placebo beetroot juice

SUMMARY:
Diseases of the heart and blood vessels, including raised blood pressure, are one of the leading causes of death worldwide. Higher intakes of dietary nitrate, found abundantly in root vegetables such as beetroot, have been shown to have health benefits including lowering blood pressure and improving the elasticity of blood vessels. Bacteria which reside in the mouth and those in the gastrointestinal tract play an important role in converting dietary nitrate to nitrite and nitric oxide (a chemical which promotes the relaxation of blood vessels). In particular, removal of oral bacteria by using antiseptic mouthwash is accompanied by an increase in blood pressure in subjects with normal blood pressure, even after consuming nitrate-rich foods. To date, very little is known about the role of these oral bacteria in the control of blood pressure, and if there are any differences in bacterial composition between individuals.

DETAILED DESCRIPTION:
Interested volunteers will be provided with an outline of the study and asked to complete a medical and lifestyle questionnaire (in person, by email or over the phone). Potentially suitable participants will be identified and asked to attend a screening session after a 12 h overnight fast (not eating during this time and only drinking water) during which the study will be explained in more detail before a consent form is signed. Anthropometric measurements will then be taken including weight, height and blood pressure. A 9 ml blood sample will also be collected on site at the Department of Food and Nutritional Sciences (Hugh Sinclair Unit of Human Nutrition). Subjects who meet the initial inclusion criteria will be invited to a further screening session during which time a dentist will check for dental diseases (e.g. current dental cavities or periodontal infection) and saliva flow rate. Volunteers without periodontal disease and with normal saliva flow will then be invited to participate in the study.

Eligible subjects will then be randomised to one of two treatments: i) up to 70 ml (the amount given will be equivalent to 3.7 mg/kg body weight) beetroot juice (James White Drinks Limited, UK) or ii) a matched volume of placebo beetroot juice (control, James White Drinks Limited, UK) to be consumed daily for 8 weeks. As drinking water is a major source of dietary nitrate, subjects will be provided with a water filter to reduce the nitrate level in their tap water for drinking and cooking during the study period. There will be a wash out period of 4 weeks between the intervention juices. In total, volunteers will be involved in the study for 20 weeks (five months).

On the day before each baseline study visit (weeks 0 and 12), volunteers will be required to fast overnight after having a low nitrate evening meal and only drinking low nitrate mineral water (Buxton mineral water), which will be provided to them, during this time. They will refrain from strenuous exercise and alcohol. On the morning of the study visit, the volunteers will be asked not to brush their teeth before they come to the clinical unit for their study visit.

When they arrive in the fasted state, the participants will be asked to provide a spot urine sample and a stool sample. Body weight and composition will be measured using the Tanita weighing scale, saliva sample and an oral bacteria sample will be collected by swabbing the tongue with a cotton swab. Volunteers will be asked to lie down for 20 minutes prior to the measurement of blood pressure and pulse wave analysis (PWA) using the Mobil-O-Graph device followed by the assessment of microvascular reactivity using Laser Doppler Imaging with iontophoresis. A blood sample of 20 ml (equivalent to just over 1 tablespoon) will then be taken before a light breakfast is provided. Volunteers will then be given a toothbrush and toothpaste to brush their teeth and asked to complete an online food frequency questionnaire (EatwellUK).

During the four-week wash-out period between interventions, participants will be instructed to avoid any beetroot juice drinks and maintain their usual dietary and lifestyle habits.

ELIGIBILITY:
Inclusion Criteria:

Male and female;

* A signed consent form;
* Blood pressure <140/90 mm Hg;
* BMI range 18.5 - 39.9 kg/m2;
* Age 18-64 years;
* Non-smoking;
* Not taking blood pressure lowering medication or using medications known to influence vascular function such as a glyceryl trinitrate (GTN) spray;
* No recent (within 3 months) or current use of antibiotics.

Exclusion criteria are:

Diagnosed with a chronic illness;

* Anaemia defined as a haemoglobin < 115 g/l for women and <130 g/l for men;
* Individuals with food allergies or allergies to medicated mouthwash or ingredients in the oral products;
* Requirements to take long-term medication active on the oral cavity including prebiotics and probiotics or have taken antibiotics within the last 3 months;
* Gingivitis diagnosis, or periodontal disease or chronic oral complaints or existing oral pathology.
* Less than four natural (enamel) buccal surfaces of upper molars available;
* Presence of fixed or removable oral appliances (e.g., dentures, orthodontic wires); xerostomia (a persistent dry mouth) diagnosis;
* Current smoker;
* Already participating in a dietary intervention study or clinical trial;
* Excessive alcohol consumption (> 14 units/wk);
* Females who are pregnant or lactating;
* Individuals not willing to give up using mouthwash or change their dental hygiene routine. Regular consumption or use of xylitol-based products such as toothpaste and chewing gum.

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 28 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2020-12-01 (Actual); Study Completion 2021-12-01 (Actual)

PRIMARY OUTCOMES:
Change in blood pressure measure | Before and after each 8 week intervention
  Systolic blood pressure, diastolic blood pressure and pulse pressure
Change in oral bacteria composition | Before and after each 8 week intervention
  Oral bacteria composition determined using next generation sequencing.

SECONDARY OUTCOMES:
Change in vascular reactivity | Before and after each 8 week intervention
  Laser Doppler Imaging with iontophoresis.
Change in Nox concentrations in serum, urine and saliva | Before and after each 8 week intervention
  Nitrate and nitrite concentrations will be determined using high performance liquid chromatography in plasma, urine and saliva. Nitric oxide will be calculated as the sum of nitrate and nitrite concentrations.
  Creatinine will be measured in the urine samples to normalise the nitrate and nitrite concentrations in urine for hydration status.
Change in gut bacteria composition | Before and after each 8 week intervention
  Stool sample will be analysed to determine composition using next generation sequencing will be used to find the differences between treatments.
Change in fasting lipid profile | Before and after each 8 week intervention
  Total cholesterol, HDL-C, and triacylglycerol will be measured using a clinical chemistry analyser. LDL-C will be calculated using the Friedewald formula.
Change in C-reactive protein | Before and after each 8 week intervention
  C-reactive protein will be measured using a clinical chemistry analyser
Change in endothelial function | Before and after each 8 week intervention
  Pulse wave analysis will be measured using Mobil-O-Graph
Change in body weight | Before and after each 8 week intervention
  Body weight will be measured using a Tanita scale
Height measurement | Before the intervention
  Height will be measured using a stadiometer
Change in body mass index | Before and after each 8 week intervention
  Body mass index will be calculated from the body weight and height measurement
Change in insulin | Before and after each 8 week intervention
  Insulin levels will be measured by ELISA
Change in glucose | Before and after each 8 week intervention
  Glucose levels will be measured using a clinical chemistry analyser
Change in insulin sensitivity | Before and after each 8 week intervention
  Glucose and insulin measurements will be used to calculate the homeostatic model assessment of insulin resistance (HOMA-IR)

CONTACTS AND LOCATIONS:
Overall Officials: Julie A Lovegrove, BSc, PhD, Principal Investigator — University of Reading
Locations (1):
- Hugh Sinclair Unit of Human Nutrition, Department of Food and Nutritional Sciences, University of Reading, Reading, Berkshire, United Kingdom